CLINICAL TRIAL: NCT05048758
Title: Vulnerability for Alcohol Use Disorder After ACE: the Role of Stress Sensitivity, Emotion Processing, Cue Reactivity and Cognitive Functions in Relapse Risk
Brief Title: Adverse Childhood Experiences in Alcohol Use Disorder
Status: Completed | Type: Observational
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GRK2350-B5-P2
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Use Disorder; Trauma, Psychological
MeSH Terms: conditions — Alcoholism; Psychological Trauma | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva (stress hormones) Blood (genotyping)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with AUD + varying levels of ACE: Individuals with alcohol use disorder (AUD) and varying levels of adverse childhood experiences (ACE)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention
  Other Names: Observational study

SUMMARY:
Adverse childhood experiences (ACE) and their relation to the development of an alcohol use disorder (AUD) will be measured with functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
The aim of this study is to examine the impact of ACE on stress sensitivity, cue-reactivity, and emotion processing in individuals with AUD at a longitudinal level. For this, participants (excluding healthy controls) from the first project (see https://clinicaltrials.gov/ct2/show/NCT03758053) will be re-examined after 2 to 2.5 years to explore the involvement of these mechanisms in relation to (long-term) relapse risk, which is a central issue in substance use disorders. Furthermore, we will investigate cognitive functions, specifically response inhibition and working memory, in the relationship between ACE and AUD. Additional participants may be recruited to mitigate sample attrition from the first project and to achieve the desired sample size. To assess cognitive functions and data from new participants in relation to relapse risk, we will perform a 3-month follow-up.

Neural correlates of stress-sensitivity, emotion processing, alcohol cue-reactivity and cognitive functions will be assessed using fMRI. Furthermore, blood and saliva samples will be used to assess biological and physiological mechanisms (e.g. salivary cortisol level or genetic markers of AUD and possible gene-environment-interactions).

The current project is interested in the extent to which ACE severity modulates neural activation in specific brain regions during the execution of fMRI paradigms as well as alcohol-related measures (e.g., craving and alcohol consumption). Of particular interest is the question whether these neural and alcohol-related measures are associated with relapse risk.

55 individuals with AUD and varying levels of ACE will be examined using interviews, questionnaires, fMRI tasks as well as saliva and blood samples. Update from 29/03/2023: the relationships of interest will be examined using a dimensional approach to the predictor variable (ACE). Thus, participants will not be divided into two groups (no or mild ACE vs. moderate to severe ACE) as originally planned, but will instead be treated as one group with varying levels of ACE. The new sample size (n = 55) is based on an updated sample size calculation for a linear regression (two-tailed) using the following input parameters: f² = 0.15 (moderate effect size), alpha error = 0.05, and power = 80%. All ethical votes and informed consents of participants will be obtained according to the declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age between 18 and 65
* Normal or correctable eyesight
* Sufficient ability to communicate with the investigators, to answer questions in oral and written form
* "Fully Informed Consent"
* "Written Informed Consent"
* Individuals with alcohol use disorder according to DSM-5 or 'heavy drinking' (alcohol intake > 40g/ more than 5 days (women) & 60g/ more than 5 days (men) and varying levels of adverse childhood experiences

Exclusion Criteria:

* Withdrawal of the declaration of consent
* Exclusion criteria for an MRI scan (pregnancy, metal implants, etc.)
* Severe internal, neurological and psychiatric comorbidities
* Pharmacotherapy with psychoactive substances within the last 14 days (except treatment with SSRI/SNRIs for at least 28 days)
* Axis-I disorder according to ICD-10 and DSM 5 (except tobacco and alcohol use disorder, substance abuse with less than 2(11) criteria according to DSM-5, mild depressive episode, adaptation disorder and specific phobia within the last 12 months)
* Positive urin drug screening (cannabis, amphetamine, opiates, benzodiazepines, cocaine)
* Withdrawal symptoms (CIWA-R > 7)
* Intoxication at time of investigation (breathalyzer > 0.3‰)
* Suicidal tendency or potential danger for others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Addiction Clinic at the Central Institute of Mental Health (Mannheim, Germany), as well as residents predominantly from the Mannheim/Heidelberg area who answered an open call to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
fMRI to assess group and within-subjects differences in task-specific brain activation patterns: Stress-sensitivity | fMRI measurement at one day only (day of fMRI experiment)
  Stress-sensitivity: Imaging Stress Task to assess neural activation patterns during mental arithmetic tasks with negative feedback
fMRI to assess group and within-subjects differences in task-specific brain activation patterns: Emotion processing | fMRI measurement at one day only (day of fMRI experiment)
  Emotion-processing: emotional face-/form-matching task to assess neural activation patters of emotion processing
fMRI to assess group and within-subjects differences in task-specific brain activation patterns: Alcohol cue-reactivity | fMRI measurement at one day only (day of fMRI experiment)
  Alcohol cue-reactivity: pictures of alcoholic beverages to assess neural alcohol-cue reactivity
fMRI to assess group differences in task-specific brain activation patterns: Response inhibition | fMRI measurement at one day only (day of fMRI experiment)
  Response inhibition: Stop Signal Task (variation of go/no-go) to assess response inhibition.
fMRI to assess group differences in task-specific brain activation patterns: Working memory | fMRI measurement at one day only (day of fMRI experiment)
  Working memory: n-back task (continuous performance) to assess working memory function.
Long-term alcohol consumption | 2 - 2.5 year follow-up after first project
  Self-report in longitudinal sample measured with the LDH interview
Short-term alcohol consumption | 3-month follow-up after current project
  Self-report in whole sample measured with the Form 90 interview

SECONDARY OUTCOMES:
Hormonal stress response using salivary cortisol level | Normal awakening response on a subject's regular week-day (0, 0.5, 8 and 14 hours after wake-up)
  Collection of saliva on a subject's regular week-day for the individual's normal cortisol awakening response and circadian rhythm (basal hypothalamic-pituitary-adrenal-function at 0, 0.5, 8 and 14 hours after wake-up).
  Cortisol awakening reaction, area under the curve and slope will therefore be calculated [nmol/L]
Hormonal stress response using salivary cortisol level | day of fMRI experiment, at -45, -22, -10 minutes before and 35, 45, 60, 75 and 90 minutes after onset of stress induction
  Time course of salivary cortisol level. Area under the curve and slope will be calculated [nmol/L]
GWAS and especially glutamatergic, serotonergic single-nucleotide polymorphisms | Blood sample at one day only (day of fMRI experiment)
  Genomic DNA using 40ml EDTA-blood

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstaedt-Klein, PhD, Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Turkmen C, Machunze N, Tan H, Gerhardt S, Kiefer F, Vollstadt-Klein S. Vulnerability for alcohol use disorder after adverse childhood experiences (AUDACE): protocol for a longitudinal fMRI study assessing neuropsychobiological risk factors for relapse. BMJ Open. 2022 Jun 30;12(6):e058645. doi: 10.1136/bmjopen-2021-058645. PMID 35772833